CLINICAL TRIAL: NCT06147752
Title: Department of Endocrinology and Diabetes, Xiamen Diabetes Institute, Fujian Province Key Laboratory of Translational Research for Diabetes, The First Affiliated Hospital of Xiamen University, School of Medicine, Xiamen, China
Brief Title: Mobile Internet Healthcare and Three Disciplines Co-management Intervention for Overweight/Obese Prediabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, zheng xin, The First Affiliated Hospital of Xiamen University, The First Affiliated Hospital of Xiamen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3502Z20224ZD1027
Record Dates: First submitted 2023-11-17; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Overweight/Obesity; Prediabetes; Weight Management
MeSH Terms: conditions — Overweight; Obesity; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile internet healthcare treatment and "three disciplines co-management" (Experimental): 100 patients who met the enrollment conditions were randomly divided into control group and intervention group by 1:1. The intervention group adopted the intervention of mobile Internet healthcare and "co-management of three disciplines" (endocrinologists, dietitians and weight managers). The three disciplines team tracked and assessed the patients' daily diet and weight changes. The duration of intervention was 6 months.
  Interventions: Behavioral: mobile internet healthcare and "co-management of three disciplines"
- Traditional diagnosis and treatment mode (Experimental): 100 patients who met the enrollment conditions were randomly divided into control group and intervention group by 1:1. The control group was treated according to the traditional mode: the diagnosis and treatment plan was formulated by the endocrinologist, and the diet education was conducted by the dietitian, and the individualized diet plan was formulated. Given a calorie-restricted diet, it is recommended to reduce daily energy intake by 500kcal on the basis of requirement. At least 150 minutes of moderate-intensity exercise per week is recommended. After the visit, the patient underwent follow-up self-weight monitoring and diet management outside the hospital.
  Interventions: Behavioral: mobile internet healthcare and "co-management of three disciplines"

INTERVENTIONS:
Behavioral: mobile internet healthcare and "co-management of three disciplines" — "co-management of three disciplines":
  Endocrinologist:
  Assess disease status and rule out secondary obesity; Identify the causes of overweight/obesity and the status and extent of associated diseases; receive patients for return visits. Timely reply to patients' questions on the mobile medical platform, and timely adjust medication plans according to changes in patients' conditions.
  Dietitians:
  Conduct diet assessment, develop personalized medicine nutrition treatment plan and provide daily real-time guidance and follow up patients' daily diet outside the hospital.
  Weight managers:
  Establish weight loss record for patients, guide the installation and use of mobile medical Application , including weight monitoring, real-time uploading of daily diet and online interactive consultation; Follow up patients' weight changes; Assist patients in making appointments for follow-up visits.

SUMMARY:
Diabetes mellitus is a chronic metabolic disease associated with a high rate of disability and mortality. Prediabetes is the intermediate stage from normal blood glucose to diabetes. Reversal of prediabetes can help reduce the incidence of related complications and reduce premature mortality. Therefore, the early treatment of prediabetes is crucial, detection and effective management of this large population in time is the key to prevent diabetes.

Overweight/obesity is one of the key risk factors leading to prediabetes and diabetes. In order to delay the progression of prediabetes and prevent related complications, weight loss is a key strategy to reverse prediabetes in overweight/obese patients. Lifestyle intervention is the first-line treatment for weight loss and is the most suitable intervention method. Although weight loss has been shown to have many metabolic benefits, it is a great challenge in the real world due to the long-term and complex of weight management.

In order to further optimize the weight loss treatment of prediabetic patients, the study apply the mobile internet intelligent healthcare big data technology, 100 overweight/obese prediabetic patients who met the enrollment conditions were randomly divided into control group and intervention group by 1:1, with 50 patients in each group. The control group was treated according to the traditional diagnosis and treatment mode, and the diagnosis and treatment plan was formulated by the endocrinologist, and the diet education was conducted by the dietitian, and the individualized diet plan was formulated. Given a calorie-restricted diet, it is recommended to reduce daily energy intake by 500kcal on the basis of requirement. At least 150 minutes of moderate-intensity exercise per week is recommended. After the visit, the patient underwent follow-up self-weight monitoring and diet management outside the hospital. The intervention group was managed by co-management of three disciplines (endocrinologists, dietitians and weight managers). The three disciplines team tracked and assessed the patients' daily diet and weight changes, and gave guidance. The duration of intervention was 6 months.

To explore the impact of the new model of mobile internet healthcare and "three disciplines co-management" on overweight/obese prediabetic patients, and whether it can improve the weight, glycemic and lipid metabolism and insulin resistance, and compare the reversal rate of prediabetes in the two groups.

DETAILED DESCRIPTION:
Sample size estimation The sample size was calculated based on the primary clinical endpoint and previous relevant clinical studies, which met 90% detection efficacy, with an a-value of 0.05 on both sides and a follow-up rate of more than 80%. 100 overweight/obese prediabetic patients were enrolled in the Department of Endocrinology and Diabetes The First Affiliated Hospital of Xiamen University.

Recruitment:

The researcher informs the patient about the study; If patients agree to participate in the study, they will need to sign an informed consent form with their doctor. The study doctor will ask and record the medical history, do physical examination, such as measuring height, weight, waist circumference, blood pressure, laboratory tests, finally determine the enrollment conditions and complete the randomized grouping. A total of 140 participants were recruited, 100 participants were finally enrolled and randomly divided into control group and intervention group according to 1:1.

Management mode:

Informed consent was signed at the first admission, and the researcher and patients were fully communicated, so that patients could realize the importance of out-of-hospital lifestyle management in reversing prediabetes. Dietitians provide detailed one-to-one guidance to each patient, using food models, pictures and other tools to guide, including food diary recording , food intake estimation, food exchange serving, nutrition label reading. Weight managers guide patients to proficiently use mobile healthcare apps, increase their attention to online communication, increase the frequency of use of online platforms for out-of-hospital care, real-time upload diet, exercise and weight monitoring indicators, respond to patient consultation in time so as to improve interaction and compliance with patients. To give full play to the effect of service management, researchers will also remind and urge patients to use apps through telephone, wechat and other ways to improve compliance.

Quality control:

1. Unified training of investigators, including program implementation, questionnaire survey, etc., to ensure unified methods in the investigation process.
2. All researcher have undergone unified training, including diagnostic standards, evaluation guidance, record norms, etc.
3. Epidata was used to build the database, and all data were entered in parallel by two people, with automatic and manual double verification.

ELIGIBILITY:
Inclusion Criteria:

①18 years≤ Age<70 years

* 5.7mmol/L≤ fasting blood glucose <6.9mmol/L

  * 7.8mmol/L≤2h blood glucose <11.0mmol/L;

    * 24Kg/m2≤BMI≤45Kg/m2

Exclusion Criteria:

* Diagnosed diabetes

  * In the past 3 months, metformin, thiazolidinedione, acarbose and weight reduction drugs were used

    * Severe infection, severe trauma or other stress

      * The weight fluctuation in the past 3 months was >5%

        * Aspartate Transaminase(AST) or Alanine Aminotransferase（ALT） increased the upper limit of 3 times the normal value; Creatinine greater than 1.5 times the upper limit of normal; Estimated Glomerular Filtration Rate（eGFR） 30 ml/min / 1.73 m2 or less

          * Serious cardiovascular and cerebrovascular disease in the past 6 months

            * Abnormal thyroid function not controlled;

              * Pregnant and breastfeeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change of weight | After 6 months of intervention, the change of weight was compared between the two groups
  Whether there was a significant difference in weight change between the intervention and control groups
Reversal rate of prediabetes | After 6 months of intervention, the reversal rate of prediabetes was compared between the two groups
  Whether there was a significant difference in the reversal rate of prediabetes between the intervention and control groups
Change of homeostasis model assessment-insulin resistance（HOMA-IR） | After 6 months of intervention, the change of HOMA-IR was compared between the two groups
  Whether there was a significant difference in HOMA-IR change between the intervention and control groups

SECONDARY OUTCOMES:
Change of BMI | After 6 months of intervention, the change of BMI was compared between the two groups
  Whether there was a significant difference in BMI change between the intervention and control groups
Change of waistline | After 6 months of intervention, the change of waistline was compared between the two groups
  Whether there was a significant difference in waistline change between the intervention and control groups
Change of serum lipid level | After 6 months of intervention, the change of serum lipid level was compared between the two groups
  Whether there was a significant difference in serum lipid level change between the intervention and control groups
Change of hepatic steatosis value | After 6 months of intervention, the change of hepatic steatosis value was compared between the two groups
  Whether there was a significant difference in hepatic steatosis value change between the intervention and control groups

CONTACTS AND LOCATIONS:
Overall Officials: xin zheng, Study Director — The First Affiliated Hospital of Xiamen University
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China